CLINICAL TRIAL: NCT05267691
Title: Basal Cell Carcinomas on Sun-protected Versus Sun-exposed Body Sites: a Clinicopathological Descriptive Study
Brief Title: Pathological Characteristics of Basal Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdulkarim Hasan, Laboratory coordinator, Al-Azhar University
Other Study IDs: AUH2201002
Record Dates: First submitted 2022-02-24; First posted 2022-03-04 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Dermatological Tumors
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sun-protected: All patients with basal cell carcinoma in a sun protected body site
  Interventions: Procedure: Excision
- sun-exposed: All patients with basal cell carcinoma in a sun exposed body site
  Interventions: Procedure: Excision

INTERVENTIONS:
Procedure: Excision — Surgical excision of the lesion and histopathology evaluation using Hematoxylin and Eosin stains

SUMMARY:
A hospital based cross-sectional study was conducted from 2017 to February 2021. Clinical history, examination and histopathological variants were collected from medical files and pathology reports. Confirmation of pathology was done in all the patients visiting skin and plastic surgery department with suspected lesions.

DETAILED DESCRIPTION:
Some cases may be tested for immunohistochemistry on the tissue block

ELIGIBILITY:
Inclusion Criteria:

* Excised lesion
* Confirmed basal cell carcinoma pathologically

Exclusion Criteria:

* Incision biopsy
* Incomplete follow up

Ages: 10 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Visiting dermatology or surgery clinics in the tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-10-20 (Estimated)

PRIMARY OUTCOMES:
Healing | 1 day
  Complete removal of the lesion

SECONDARY OUTCOMES:
Recurrence | 1 year
  Occurrence of recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Abdulkarim Hasan, Principal Investigator — Al-Azhar University
Locations (1):
- Abdulkarim Hasan, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No